CLINICAL TRIAL: NCT06158477
Title: An Open-label Multicenter, Phase I Clinical Study to Evaluate the Safety, Tolerability, and Pharmacokinetic Characteristics of JYP0035 Capsule Monotherapy in Patients With Advanced Solid Tumors
Brief Title: A Clinical Trial Evaluating JYP0035 Capsule Monotherapy in Patients With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Chengdu JOYO pharma Co., Ltd. (Industry)
Collaborators: Guangzhou JOYO Pharma Co., Ltd (Industry)
Responsible Party: Sponsor
Organization: Guangzhou JOYO Pharma Co., Ltd (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: JYP0035M101
Record Dates: First submitted 2023-11-28; First posted 2023-12-06 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- JYP0035 monotherapy dose-escalation group (Experimental): PART-1 Single Dose Escalation Group
  Interventions: Drug: JYP0035 Experimental Drug Treatment
- JYP0035 monotherapy dose-expansion group (Experimental): PART-2 JYP0035 Monotherapy Dose Expansion Group
  Interventions: Drug: JYP0035 Experimental Drug Treatment

INTERVENTIONS:
Drug: JYP0035 Experimental Drug Treatment — Single dose intervention

SUMMARY:
The goal of this Phase I clinical trial is to evaluate the safety, tolerability, and pharmacokinetic characteristics of the JYP0035 capsule in patients with advanced solid tumors. The main questions it aims to answer are:

* What is the safety profile of JYP0035 when administered to these patients?
* How does JYP0035 capsule behave in the body pharmacokinetically?

Participants will:

* Receive escalating doses of JYP0035 capsule during the dose-escalation phase (PART-1).
* Continue with the identified dose in the dose-expansion phase (PART-2).

As this is a single-arm study, there is no comparison group.

ELIGIBILITY:
Inclusion Criteria:

* Patients voluntarily participate in the clinical trial and sign the informed consent form
* Age 18 years and above (inclusive), and below 75 years of age (inclusive), with no gender restrictions
* ECOG(Eastern Cooperative Oncology Group)performance status of 0 or 1
* Expected survival time of ≥3 months
* During the screening period, female patients of childbearing potential must have a negative serum pregnancy test within 7 days prior to administration of the study drug
* Participants agree to use reliable contraception methods from signing the informed consent form until 6 months after the last dose of the study drug. This includes, but is not limited to: abstinence, vasectomy in males, female sterilization, effective intrauterine devices, and effective contraceptive medications

Exclusion Criteria:

* Participants have not recovered to normal or ≤ Grade 1 from any adverse events and/or complications caused by any previous treatments before the first administration of the study drug, excluding hair loss and pigmentation
* Patients with imaging (CT or MRI) showing tumor invasion into major blood vessels (such as the aorta, pulmonary arteries and veins, vena cava, etc.)
* Patients who have had clinically significant cardiovascular or cerebrovascular diseases within 6 months before the first administration, which, in the investigator's judgment, may interfere with the patient's full participation in the study; atrial fibrillation; clinically significant supraventricular or ventricular arrhythmias requiring treatment or intervention
* Patients who had history of type 1 diabetes, type 2 diabetes, or gestational diabetes
* Individuals with other malignancies or with a history of other malignant tumors
* Individuals with a history of severe allergies, or who are allergic to any active or inactive ingredients of the study drug
* Pregnant or breastfeeding patients
* Researchers consider participants unsuitable for this clinical study due to any clinical or laboratory abnormalities or other reasons

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Assess the adverse event rate of this clinical trial | From 8 weeks after the first administration up to week 52
  Grading the adverse events using National Cancer Institute - Common Terminology Criteria for Adverse Events(NCI-CTCAE)version 5.0.

SECONDARY OUTCOMES:
Assess Area Under the Curve(AUC) | From 8 weeks after the first administration up to week 52
  Area under the plasma concentration-time curve from zero to infinity

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No